CLINICAL TRIAL: NCT04719156
Title: Evaluation of Intraoperative Tumor Margin Identification with Fluorescent Dye Imaging
Brief Title: Fluorescent Intra-operative Tumor Margin Examination
Acronym: ICGTM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kurt Weiss (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor-Investigator, Kurt Weiss, Principal Investigator, Associate Professor, Director, Musculoskeletal Oncology Lab, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY19110051
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Indocyanine Green; Injections

STUDY DESIGN:
Intervention Model Description: Patients with suspected sarcoma tumors.
Masking Description: Operating surgeon will be blinded to ICG Images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ICG use followed by SPY-PHI imaging. (Other): Participants will be injected with 2.0mg/kg of ICG dye to access tumor margin using Stryker SPY imaging technology.
  Interventions: Drug: Indocyanine green solution administered at 2.0mg/kg.; Device: Stryker SPY-PHI Imaging Device

INTERVENTIONS:
Drug: Indocyanine green solution administered at 2.0mg/kg. — Dosing of ICG to be administered at 2.0mg/kg, two hours prior to surgery.
  Other Names: Indocyanine Green for Injection
Device: Stryker SPY-PHI Imaging Device — The SPY-PHI system is used with the ICG dye to provide fluorescence images.
  Other Names: Stryker SPY portable Imaging System

SUMMARY:
Tumor margin confirmation is important to confirming appropriate disease excision. Current standard of care is to take select margin samples to pathology for intra-operative readings. However, this is expensive, time consuming, and only assesses the margin contained within the specific sample. In prior work the investigators have determined that indocyanine green (ICG) is highly specific to the tumor bed when injected shortly before surgery. The investigators hypothesize that ICG will be able to accurately identify residual positive tumor margins during sarcoma excision procedures.

DETAILED DESCRIPTION:
Experimental Design:

1. A physician investigator will obtain consent during the pre-operative appointment. Study team members may assist with the discussion.
2. Upon arrival to the pre-operative area 2 hours prior to surgery, the participant will be injected with 2.0 mg/kg ICG (Indocyanine Green Dye) as per standard protocol: during regular pre-operative work-up, during which a standard of care IV is inserted. The PI or resident physician will administer the injection.
3. The participant will undergo the tumor removal surgery as planned pre-operatively.

   To assess the accuracy and precision of ICG dye localization within tumor, not non-tumor, a small sample of tumor and a small sample of native tissue will be obtained for microscopy analysis (ICG fluorescence is possible on slides following frozen sectioning) 30 seconds, no intra-operative delay.
4. Once the tumor is removed to the satisfaction of the surgeon, ICG Angiography (SPY PHI) will be performed to detect any residual signal, 2-3 minutes, no re-draping required.

   The surgeon will complete a "feedback sheet" that assesses if the tumor was completely excised (or an intentional positive margin was left).
5. The operative surgeon will be blinded to the angiography result. ICG Angiography will be performed by the resident or surgical staff, without surgeon involvement. No study team members are blinded.
6. The dose that will be administered 2.0 mg/Kg IC. Doses are being based on measurements on post-washout signal (or the remaining signal after the dye is metabolized). Weight based dosing is therefore far more important. The proposed dosing is not close to the LD50 (median lethal dose) of ICG and no side effects are anticipated with the increased dose.
7. The Stryker team will be perform an in-service for SPY PHI ( SPY portable hand held imaging device) for all OR staff members, and individual demonstrations for each service resident will be performed. The device is very simple to use and no active measurements need to be made. No extended anesthesia will be required.
8. The participant will be monitored for recurrence, which will be compared with ICG angiography findings intra-operatively.
9. Study efficacy will be evaluated every 6 months, as early-termination and clinical translation will be indicated should accuracy be proven in compliance with IRB (Institutional Review Board) "do no harm" rules.
10. Radiographs, that are completed post operatively during the standard of care visit, will be reviewed for this research.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 with a primary musculoskeletal tumor that has been indicated for surgical excision by a fellowship trained orthopaedic oncologist.
* Surgical consent was obtained prior to research consent.
* Patients with a biopsy-confirmed primary soft tissue or bone tumor that has not been previously excised and has a known risk of local or remote recurrence.

Exclusion Criteria:

* Patients below the age of 18
* Pregnancy, breast feeding
* Patients with a history of anaphylactic reaction to contrast media or fluorescein allergy
* Prior surgery local to the mass being excised
* Non- or minimally-recurrent masses (i.e. osteochondroma)
* Dialysis, renal failure, uremia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence as predicted by the surgeon vs. identified with SPY. | During surgery for tumor removal
  The proportion of tumors declared "completely removed" by the surgeon that recur locally will be compared those with SPY-identified residual disease.

SECONDARY OUTCOMES:
Comparison of ICG angiography with pathologic evaluation | Over a two year follow up period
  The ICG signal accessed at the time of surgery, will be compared with final anatomic pathology in order to discern its degree of accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Weiss, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No